CLINICAL TRIAL: NCT05792358
Title: Wet Cupping Therapy in Ankylosing Spondylitis: a Multicenter Randomised Controlled Trial
Brief Title: Wet Cupping Therapy in Ankylosing Spondylitis
Status: Enrolling by invitation | Phase: Not Applicable | Type: Interventional
Sponsor: Karabuk University (Other)
Responsible Party: Principal Investigator, SULEYMAN ERSOY, Head of the complementary medicine department, Karabuk University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: SBU177
Record Dates: First submitted 2023-03-07; First posted 2023-03-31 (Actual); Last update posted 2024-07-25 (Actual); Status verified 2024-07

CONDITIONS: Ankylosing Spondylitis
Keywords: Ankylosing Spondylitis; Wet cupping therapy; Basfi; Basdai; Vas
MeSH Terms: conditions — Spondylitis, Ankylosing

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Wet cupping arm (Experimental): This arm is the interventiom group and will receive three consecutive sessions of wet cupping therapy once a month.
  Interventions: Procedure: wet cupping therapy
- Control arm (No Intervention): This arm is the control group and will not receive any intervention other than the routine medications

INTERVENTIONS:
Procedure: wet cupping therapy — wet cupping therapy will be applied to participants in this arm for three sessions once a month
  Arms: Wet cupping arm

SUMMARY:
This study evaluates the efficacy of wet cupping therapy in patients with ankylosing spondylitis.Wet cupping therapy will be applied to half of the patients plus routine pharmaceutical treatment while the other half will receive only pharmaceutics

DETAILED DESCRIPTION:
In addition to the medical treatment, WCT will be applied once a month, 3 times (Day 0, 30, 60) to the intervention group whereas the control group will not receive any intervention. The BASFI, BASDAI, VAS and Schober test will be applied to both groups at 0 and 3 months.

ELIGIBILITY:
Inclusion Criteria:

Clinical diagnosis of ankylosing spondylitis 18-65 years of age Consent to participate

Exclusion Criteria:

Any ongoing medical treatment other than NSAIDs Pregnancy At least one contraindication to WCT that was detected in subject's history or in the routine blood examinations prior to enrollment (Hgb <9.5; INR> 1.2; history of hemophobia, bleeding disorder, malignant disorder).

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2023-02-01 (Actual); Primary Completion 2025-07-01 (Estimated); Study Completion 2025-12-01 (Estimated)

PRIMARY OUTCOMES:
BASFI | At 0 and 3 months
  Change in the scores of The Bath Ankylosing Spondylitis Functional Index
BASDAI | At 0 and 3 months
  Change in the scores of The Bath Ankylosing Spondylitis Disease Activity Index
VAS | At 0 and 3 months
  Change in the scores of Visual Analogue Scale

SECONDARY OUTCOMES:
Schober | At 0 and 3 months
  Change in the scores of Modified Schober Test

CONTACTS AND LOCATIONS:
Locations (1):
- Karabuk University, Karabük, Turkey (Türkiye)